CLINICAL TRIAL: NCT05319496
Title: Intermittently Scanned CGM Versus Usual Care With Diabetes Education and Feedback, in Adults With Non-Insulin Dependent Type 2 Diabetes (iCUDE): A Randomized Trial
Brief Title: isCGM With Education and Feedback for Non-Insulin Dependent Type 2 Diabetes
Acronym: iCUDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Epidemiology Coordinating and Research Centre, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00119503
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: continuous glucose monitoring; flash glucose monitoring; intermittently scanned continuous glucose monitoring; CGM; non-insulin dependent diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- isCGM with education and feedback (Experimental): Intervention subjects will receive three isCGM sensors (FreeStyle Libre 2, Abbott Laboratories) for use over weeks 1-6. They will have encounters with a diabetes educator for individualized education and coaching during weeks 1-2 and 5-6.
  Interventions: Device: Intermittently scanned continuous glucose monitor (isCGM); Behavioral: Education and coaching
- Enhanced usual care with education and feedback only (Active Comparator): Enhanced usual care subjects will receive two encounters with a diabetes educator for individualized education and coaching, during weeks 1-2 and 5-6. They will not be provided with isCGM sensors.
  Interventions: Behavioral: Education and coaching

INTERVENTIONS:
Device: Intermittently scanned continuous glucose monitor (isCGM) — A wearable sensor the size of 2 stacked quarters, that allows individuals to "scan" their glucose levels on demand. No fingerstick is required. The device measure interstitial glucose through a filament that is inserted under the skin. The application process is painless, and each sensor lasts 90 days. Sensors can be scanned with certain smart phones. This device is marketed as the FreeStyle Libre 2 glucometer (Abbott Laboratories, IL).
  Other Names: Flash glucose monitor
  Arms: isCGM with education and feedback
Behavioral: Education and coaching — Two encounters with a certified diabetes educator, who will assess lifestyle and medications, and provide individualized advice on diet, physical activity, and medication changes to improve glycemic control.

SUMMARY:
Glycemic control is an important for adults with diabetes. Self-monitoring of glucose can help adults with type 2 diabetes (T2DM) meet their glucose targets. Continuous glucose monitoring (CGM), an alternative to traditional capillary (finger-stick) blood glucose, uses a wearable sensor that continuously measures glucose levels under the skin. With intermittently scanned CGM (isCGM), patients scanning the sensor to obtain readings. isCGM is painless, provides information on glucose trends, and has improves patient satisfaction.

Most adults with diabetes are not on insulin. Yet, the effectiveness of CGM is not well studied in this population. In this randomized trial, we are looking for adults with type 2 diabetes, who need further blood glucose lowering (HbA1c > 7.0%), who are not yet on insulin. Participants randomized to the treatment group (50%) will receive isCGM with individual coaching; those in the the enhanced usual care group (50%) will receive diabetes coaching only. The intervention will feature three FreeStyle Libre 2 (Abbott Laboratories, IL) sensors (6 weeks), and is intended to be affordable and applicable to a wide range of adults with diabetes under real world conditions.

DETAILED DESCRIPTION:
Objective: To evaluate the effectiveness of intermittently scanned continuous glucose monitoring (isCGM) with education and feedback on glycemic control at 12 weeks, in adults with type 2 diabetes and uncontrolled HbA1c (> 7.0%) not on insulin therapy.

Background: Continuous glucose monitoring (CGM) has been shown to reduce hypoglycemia in adults on insulin. The effectiveness of CGM in adults with type 2 diabetes not on insulin therapy has not been well studied. We hypothesize that isCGM linked to structured education - specifically one-on-one review and feedback of glucose values with a diabetes educator - can improve HbA1c via a combination of improved lifestyle choices and accelerated medication intensification, in adults with earlier T2DM. To test this hypothesis, we propose a randomized controlled trial of isCGM + structured education, versus enhanced usual care with structured education only.

Methods: Open-label, 12-week, single-center randomized controlled trial. Included adults will be randomized 1:1 to intervention or enhanced usual care. Intervention participants will receive three FreeStyle Libre 2 (Abbott Laboratories, IL) isCGM sensors to be applied over weeks 1-6. Diabetes education and coaching will be provided at the beginning and end of the sensor period. The control group will receive diabetes education and coaching during weeks 1-2 and 5-6, but not the isCGM sensors. The primary outcome (HbA1c change from baseline) will be measured by venous blood draw at 12 weeks. Participants will be asked to complete patient-reported outcome instruments for secondary outcomes, e.g.: diabetes self-empowerment, diet, and physical activity - at baseline, 6 weeks, and 12 weeks.

Significance: This trial will examine the effectiveness of scheduled, intermittent use of isCGM sensors for type 2 diabetes, when combined with education and feedback. The intervention is designed to be affordable and applicable to a wide range of adults with diabetes, and may have significant implications for the use of isCGM.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years with type 2 diabetes.
* HbA1c > 7.0% within the last 6 months.
* Non-insulin therapy.
* Able to attend two in-person study visits.
* English-speaking.
* Community-dwelling
* In possession of a cell phone capable of accessing the internet and receiving FreeStyle Libre 2 sensor readings
* Has a primary care provider who has been in contact with the patient for diabetes in the last 12 months.

Exclusion Criteria:

* Type 1 diabetes or diabetes clearly identified as having monogenetic etiology (e.g.: MODY).
* Steroid-induced diabetes if steroid use is on-going or most recently taken within the last 3 months.
* Pregnancy; plans to become pregnant within 6 months; breast-feeding.
* Any use of insulin in the previous year.
* Current or previous use of isCGM or rtCGM within the last 6 months.
* Cognitive dysfunction (SPMSQ score >= 5).
* Symptoms of acute metabolic decompensation (extreme thirst, high urinary output, and weight loss, accompanied by acute fatigue or dyspnea).
* Any terminal condition that would limit life expectancy to < 1 year.
* Inability to use isCGM (e.g.: afraid of the device).
* Inability to be reached by telephone.
* Concurrent participation in a different diabetes-related trial.
* Has not already received two doses of a Health Canada-approved vaccine against SARS-CoV-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 12 weeks
  Change in HbA1c assessed by venous blood draw, compared to baseline.

SECONDARY OUTCOMES:
Diabetes treatment satisfaction | 6 weeks and 12 weeks
  Difference in Diabetes Treatment Satisfaction Questionnaire (DTSQ) score from baseline (DTSQs scores range 0-36, higher indicating better treatment satisfaction); DTSQc "change" score at 6 weeks.
Diabetes self-care empowerment | 6 weeks and 12 weeks
  Change in Diabetes Empowerment Scale - Short Form (DES-SF) score from baseline. DES-SF score ranges 1-5, higher scores indicating greater self-care empowerment.
Diabetes-related distress | 6 weeks and 12 weeks
  Change in Problem Areas in Diabetes Questionnaire (PAID) score from baseline. PAID score ranges 0-100, a score above 40 indicates severe diabetes distress.
Healthy diet | 6 weeks and 12 weeks
  Change in UK Diabetes and Diet Questionnaire (UKDDQ) score from baseline. UKDDQ score ranges 0-5 with higher scores indicating more healthy dietary choices.
Physical activity | 6 weeks and 12 weeks
  Change in International Physical Activity Questionnaire (IPAQ) short form score. IPAQ score estimates total metabolic equivalent-minutes per week, with higher scores indicating more a more physically active individual.
Health-related quality of life | 6 weeks and 12 weeks
  Change in Euroqol EQ-5D-5L health utility score from baseline. EQ-5D scores range from 0-100, with 100 indicating a state of perfect health.
Emergency department visits | 12 weeks
  Number of emergency department visits during the 12-week trial period.
Hospital admissions | 12 weeks
  Number of hospital admissions during the 12-week trial period.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Lau, MD/PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital / Kaye Edmonton Clinic, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olu-Jordan I, Singh P, Zhang JR, Yeung RO, Manca DP, Perry T, Rahim G, Hagen E, Lau D. The Effects of Continuous Glucose Monitoring on Patient-reported Outcomes in Adults with Non-Insulin-dependent Type 2 Diabetes: A Randomized Controlled Trial. Can J Diabetes. 2025 Oct 27:S1499-2671(25)00354-5. doi: 10.1016/j.jcjd.2025.10.174. Online ahead of print. PMID 41161400

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT05319496/Prot_SAP_ICF_001.pdf